CLINICAL TRIAL: NCT06420050
Title: Testing a Novel Instagram Intervention for Heavy Alcohol Use: A Randomized Controlled
Brief Title: Testing a Novel Instagram Intervention for Heavy Alcohol Use
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Emily Grekin (Other)
Responsible Party: Sponsor-Investigator, Emily Grekin, Associate Chair, Wayne State University
Organization: Wayne State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-23-11-6344
Record Dates: First submitted 2024-04-10; First posted 2024-05-17 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Heavy Drinking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instagram Intervention (Experimental)
  Interventions: Behavioral: Instagram Intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Instagram Intervention — The intervention consists of a study Instagram page, which will post intervention content every day for 42 days.
  Arms: Instagram Intervention

SUMMARY:
This project aims to test the efficacy of an Instagram-based intervention for reducing heavy alcohol use. More specifically, the investigators will use a randomized controlled design to analyze differences in alcohol use and alcohol-related outcomes (e.g., alcohol-related consequences, etc.) as well as differences in the use of protective behavioral strategies and mindfulness practices. Participants (80 Prolific users who report binge drinking) will be randomly assigned to 1 of 3 conditions: intervention or control. Those who are randomized to the intervention condition will be invited to follow study Instagram pages, and those who are randomized to the control condition will be invited to complete the assessments only. The investigators hypothesize that there will be greater reductions in alcohol use, frequency, and consequences and greater frequency of use of mindfulness exercises and protective behavioral strategies among those in the intervention condition as compared to those in the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-30
* Report regular Instagram usage (i.e., at least a few times a week)
* Report having met the NIAAA's criteria for a binge-drinking episode (4+ drinks in a sitting for cisgender women, 5+ drinks in a sitting for all other genders) at least twice a month for the past three month

Exclusion Criteria:

* No exclusion criteria

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-22 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Frequency of Past-month Alcohol Use Using the Computer-Administered Timeline Follow-Back | Given pre-intervention and at 10-week follow-up
  The investigators will analyze differences in the amount of days spent drinking.
Change in Quantity of Past-month Alcohol Use Using the Computer-Administered Timeline Follow-Back | Given pre-intervention and at 10-week follow-up
  The investigators will analyze differences in amount of past-month alcohol use and the amount of past-month binge-drinking episodes.

SECONDARY OUTCOMES:
Change in Frequency of Protective Behavioral Strategy Use Using the Protective Drinking Practices Scale | Given pre-intervention and at 10-week follow-up
  The investigators will analyze the difference in frequency of recent protective behavioral strategy use using the Protective Drinking Practices Scale (minimum score = 20, maximum score = 120, and higher scores indicate a better outcome).
Change in the Amount of Recent Alcohol Consequences Using the Brief Young Adult Consequences Scale | Given pre-intervention and at 10-week follow-up
  The investigators will analyze the difference in amount of consequences related to alcohol use using the Brief Young Adult Consequences Scale (minimum score = 0, maximum score = 24, and higher scores indicate a worse outcome).
Change in Frequency of Mindfulness Practice Use Using the Mindfulness Awareness Scale | Given pre-intervention and at 10-week follow-up
  The investigators will analyze the difference in frequency of use of mindfulness practices using the Mindfulness Awareness Scale (minimum score = 15, maximum score = 90, and higher scores indicate a better outcome).
Change in Readiness to Change Drinking Behavior Using the Readiness to Change Questionnaire | Given pre-intervention and at 10-week follow-up
  The investigators will analyze the difference in reported readiness to change drinking behavior using the Readiness to Change Questionnaire (minimum score = 12, maximum score = 84, and higher scores indicate a better outcome).
Participant Subjective Reactions Using Likert Scales | Given at 10-week follow-up
  The investigators will ask participants to rate the intervention content on acceptability dimensions created specifically for this study (i.e., relevance, empathy, interest, helpfulness, respectfulness, personalization). On a given domain, minimum score = 1, maximum score = 5, and higher scores indicate better outcomes.
Participant Subjective Reactions Using Simple Yes/No Questions | Given at 10-week follow-up
  The investigators will ask participants to rate how the intervention has qualitatively impacted them using simple yes/no questions (i.e., if they remember seeing certain posts, if the posts made them think about their drinking, affected their sense of community, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT06420050/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT06420050/ICF_001.pdf